CLINICAL TRIAL: NCT00575601
Title: Effects of Simvastatin on Biochemical Parameters and Outcome of IVF-ICSI in Pcos Patients : A Prospective Randomized Double Blind Placebo Controlled Trial
Brief Title: Effects of Simvastatin on Biochemical Parameters and Outcome of IVF-ICSI in Pcos Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Akabr Fotouhi, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 850-39-4796
Record Dates: First submitted 2007-12-15; First posted 2007-12-18 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-06

CONDITIONS: Polycystic Ovary Syndrome
Keywords: pco; simvastatin; ivf; embryo transfer
MeSH Terms: conditions — Polycystic Ovary Syndrome; Long Qt Syndrome 3 | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: SIMVASTATIN
- B (Placebo Comparator)
  Interventions: Drug: SIMVASTATIN

INTERVENTIONS:
Drug: SIMVASTATIN — 20 mg/day,po,for two months until the day of hCG injection placebo pills as like as simvastatin will be used

SUMMARY:
The purpose of this study is to determine whether simvastatin is effective in the improvement of IVF-ICSI outcome in Pcos patients.

DETAILED DESCRIPTION:
simvastatin reduces cardiovascular risks by improving hypercholesterolemia, reducing vascular smooth muscle proliferation, ameliorating inflammation, limiting theca-interstitial proliferation & decreasing steroidogenesis (production of progesterone & testosterone).Polycystic ovary syndrome (pcos) is associated with increased cardiovascular risks and is characterized by ovarian theca-interstitial hyperplasia& hyperandrogenism .This study will test the hypothesis that simvastatin improves biochemical parameters& IVF-ICSI outcome in Pcos patients.

ELIGIBILITY:
Inclusion Criteria:

* Pcos patients
* Age <40 years
* FSH<10 IU/L

Exclusion Criteria:

* Endometriosis grade 3 &4
* History of tubal surgery
* Hydrosalpinx
* History of mellitis diabetes

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-08; Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
ivf-et outcomes | 14-20 days

SECONDARY OUTCOMES:
Biochemical parameters baseline and 8weeks Biochemical parameters | baseline and 8weeks

CONTACTS AND LOCATIONS:
Overall Officials: batool hossein rashidi, MD, Study Chair — Tehran University of Medical Sciences
Locations (1):
- Imam Khomeiny Hospital, Tehran, Iran

REFERENCES:
- [Derived] Xiong T, Fraison E, Kolibianaki E, Costello MF, Venetis C, Kostova EB. Statins for women with polycystic ovary syndrome not actively trying to conceive. Cochrane Database Syst Rev. 2023 Jul 18;7(7):CD008565. doi: 10.1002/14651858.CD008565.pub3. PMID 37462232
- [Derived] Rashidi B, Abediasl J, Tehraninejad E, Rahmanpour H, Sills ES. Simvastatin effects on androgens, inflammatory mediators, and endogenous pituitary gonadotropins among patients with PCOS undergoing IVF: results from a prospective, randomized, placebo-controlled clinical trial. J Investig Med. 2011 Aug;59(6):912-6. doi: 10.2310/JIM.0b013e31821bfd9c. PMID 21527854